CLINICAL TRIAL: NCT00330161
Title: Phase II Evaluation of Suberoylanilide Hydroxamic Acid (NSC 701852) in Patients With Advanced Prostate Cancer That Has Progressed on One Prior Chemotherapy
Brief Title: Vorinostat in Treating Patients With Progressive Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03067; NCI-2012-03067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2005.127 (Other: University of Michigan); 6862 (Other: CTEP); N01CM62206 (NIH); N01CM62201 (NIH); U01CA062491 (NIH); P30CA046592 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral vorinostat (SAHA) once daily on days 1-21. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) after 4 courses receive an additional 3 courses. All other patients may continue treatment in the absence of disease progression or unacceptable toxicity.
  Blood samples are taken on day 15 of course 1, day 1 of course 2, during the last week of course 4, and at completion of study treatment. Blood is examined for interleukin (IL)-6, IL-6 receptor, and gp130 levels.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with progressive metastatic prostate cancer. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of oral SAHA in patients with castrate metastatic prostate cancer who have progressed on one prior chemotherapy, as measured by the proportion of patients not progressed at 6 months.

SECONDARY OBJECTIVES:

I. To evaluate the safety of oral SAHA in patients with castrate metastatic prostate cancer who have progressed on one prior chemotherapy.

II. To assess the objective response rate of oral SAHA in patients with measurable disease when present.

III. To assess the rate of PSA decline of >= 50%. IV. To assess progression free and median survival in patients with castrate metastatic prostate cancer who have progressed on one prior chemotherapy.

V. To evaluate pre and post-treatment tumor biopsies when available for the presence of changes in the expression of AR and Hsp90 client proteins, Thioredoxin, Thioredoxin Binding Protein, HDAC 3 (class I), HDAC 7 (class II), EZH2 and p21 expression.

VI. To determine the effects of oral SAHA on IL-6, soluble IL-6 receptor and soluble gp130 levels in the blood.

VII. To determine the accumulation and biodistribution of 18FDHT and correlate these findings with standard FDG PET, radionuclide bone scan, CT and/or MRI scans, as well as 18FDHT pharmacokinetics and tumor tissue staining for androgen receptor (AR) and Hsp90 client proteins (this applies only to patients at MSKCC under a separate protocol #00-095).

OUTLINE: This is a multicenter study.

Patients receive oral vorinostat (SAHA) once daily on days 1-21. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) after 4 courses receive an additional 3 courses. All other patients may continue treatment in the absence of disease progression or unacceptable toxicity.

Blood samples are taken on day 15 of course 1, day 1 of course 2, during the last week of course 4, and at completion of study treatment. Blood is examined for interleukin (IL)-6, IL-6 receptor, and gp130 levels.

After completion of study treatment, patients are followed periodically for survival.

ELIGIBILITY:
Inclusion Criteria:

* A histologic or cytologic diagnosis of prostate cancer
* Metastatic prostate cancer with measurable and/or bony disease that has progressed despite androgen deprivation therapy and one prior chemotherapy for castrate metastatic disease; all patients must have PSA progression defined as:

  * At least 2 rises in PSA to be documented over a reference value (measure 1); the first rising PSA (measure 2) must be taken at least 7 days after the reference value; a third confirmatory PSA measure is required to be greater than the second measure and must be obtained at least 7 days after the 2nd measure; if this is not the case, a fourth PSA is required to be taken and be greater then the 2nd measure
* All patients must have a minimum PSA of >= 5 ng/ml
* ECOG performance status of 0-2
* Testosterone < 50 ng/dL; patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy
* No investigational or commercial agents (other than LHRH analogue) or therapies including other hormonal agents such as megestrol acetate (unless low dose given for hot flashes), antiandrogens or herbal medications may be administered with the intent to treat the patient's malignancy
* Four weeks must have elapsed since major surgery
* Prior radiotherapy is allowed as long as the bone marrow function is adequate and at least 4 weeks has elapsed since completion of radiation; no prior radiopharmaceuticals are allowed
* Life expectancy of greater than 6 months
* Ability to understand and the willingness to sign a written informed consent document that is approved by the Institutional Human Investigation Committee (HIC)
* Patients must have normal organ and marrow function as defined below obtained within two weeks from treatment initiation:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Serum creatinine < 2 mg/DL
* Total bilirubin within normal institutional limits
* AST/ALT =< 2.5 X institutional upper limit of normal
* Patients must be willing to provide blood samples for the correlative studies and consent to providing paraffin blocks/slides from primary prostate cancer or other prior diagnostic samples; fresh tissue sample donation is optional
* The effects of SAHA on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because HDAC inhibitors are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Patients with treated and controlled epidural disease are permitted into the study

Exclusion Criteria:

* Significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months)
* Patients on Valproic Acid (a histone deacetylase inhibitor) must have stopped taking it at least 2 weeks prior to registration
* Oral anti-androgens must be stopped; no washout period is necessary prior to enrollment if anti-androgens were used as second line therapy and not as part of combined androgen deprivation; in the unlikely case that a patient may have continued on antiandrogen therapy as part of combined androgen deprivation and has never had antiandrogen withdrawal despite progression on combined androgen deprivation then a washout period will be needed (4 weeks for flutamide and 6 weeks for bicalutamide or nilutamide) prior to study enrollment
* Patients who have developed progression as defined in this protocol on stable doses of oral corticosteroids are eligible; the steroids may be continued
* No "currently active" second malignancy other than non-melanoma skin cancer; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be with no evidence of disease
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, brain scans will not be required as part of the pre-study workup
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients with history of HIV receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SAHA; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients with the following history or clinical findings require ADDITIONAL diagnostic TESTING:

  * Patients who require diuretics for reasons other than hypertension, digoxin for reasons other than atrial fibrillation, or patients with a history of mild to moderate congestive heart failure
  * Patients with the following EKG results:

    * Significant q waves (greater than 3 mm or greater than 1/3 the height of the QRS complex
    * ST elevation or depressions of greater than 2 mm that are not attributable to hypertension strain
    * The absence of a regular sinus rhythm
    * The presence of a bundle block
  * ADDITIONAL TESTING: (if required)

    * Radionuclide angiocardiography (RNCA): Patients can be treated if the ejection fraction is > 45% and there is no evidence of ventricular aneurysm or other abnormal wall motion; patients with an ejection fraction < 45% on RNCA, with a worrisome but nonexclusive cardiovascular history, or an abnormal ECG as described above should also have a thallium stress test

      * STRESS TEST RESULTS:

        * Reversible defect - Exclude
        * Fixed defect alone - Include

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-03; Primary Completion 2009-09 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 medical centers between May 2006 and February 2007.
Period: Overall Study
Arm/Group | Treatment (Vorinostat)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 29 patients enrolled, only 27 were analyzed. Two patients were deemed ineligible after treatment started and they were excluded from all analysis except adverse event collection.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years]
  Age | 68 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who do Not Demonstrate Disease Progression
Description: Fisher's Exact Test will be used.
Time Frame: At 6 months
Population: The primary objective was to determine the number of patients wtih progression-free survival at 6 months. Unfortunately all eligible patients were off therapy before the 6 month time point. 13 (48%) were removed due to progression, 11 (41%) secondary to toxicity, and 3 (11%) for other reasons.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Toxicity
Description: The percentage of eligible participants that experience grade 3 or 4 toxicities.
Time Frame: Up to 3 years
Population: Of the 29 patients enrolled, 2 were deemed ineligible after treatment and therefore excluded from outcome analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 27
percentage of participants | 48

3. Secondary Outcome: Rate of PSA Decline
Description: Rate of Prostate Specific Antigen (PSA) decline of greater than or equal to 50%.
Time Frame: Up to 3 years
Population: No PSA declines of greater than or equal to 50% were observed, therefore the rate could not be determined.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Median time to progression was determined.
Time Frame: From the start of treatment to time of progression, assessed up to 3 years
Population: Of the 29 patients enrolled, two patients were deemed ineligible after treatment and therefore excluded from analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 27
months | 2.8 [0.5 to 5.3]

5. Secondary Outcome: Median Survival
Description: Median overall survival.
Time Frame: Up to 3 years
Population: Of the 29 patients enrolled, two patients were deemed ineligible after treatment and therefore excluded from analysis. Of the 27 patients analyzed, one patient was censored with an outlying overall survival of 15.1 months.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 26
months | 11.7 [2.3 to 14]

6. Secondary Outcome: Objective Response Rate
Description: Percentage of participants that obtain the best objective response, stable disease.
Time Frame: Up to 3 years
Population: Of the 29 patients enrolled, two patients were deemed ineligible after treatment and therefore excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 27
percentage of participants | 7

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were reported that occurred within 30 days of the last dose of study drug.
Description: All patients were evaluable for toxicity from the time of their first treatment with SAHA.
Arm/Group | Treatment (Vorinostat)
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=29)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage Urinary Tract (Renal and urinary disorders) | 1 (1)
Infection, Bone (Osteomyelitis) (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=29)
Abdominal Distention (Gastrointestinal disorders) | 2 (2)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 (18)
Alanine Aminotransferase Increased (Investigations) | 5 (5)
Alkaline Phosphatase Increased (Investigations) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 21 (36)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 6 (14)
Bladder Hemorrhage (Renal and urinary disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 11 (18)
Dry Mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema Limbs (General disorders) | 2 (3)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (2)
Fatigue (General disorders) | 25 (57)
Fever (General disorders) | 3 (3)
Hearing Loss (Ear and labyrinth disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 11 (19)
Hot Flashes (Vascular disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 3 (5)
Hypersensitivity (General disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
INR Increased (Investigations) | 3 (28)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Leukopenia (White Blood Cells Decreased) (Investigations) | 4 (12)
Lymphopenia (Investigations) | 3 (4)
Mucositis Oral (Gastrointestinal disorders) | 3 (4)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Platelet Count Decreased (Investigations) | 15 (20)
Taste Alteration (Nervous system disorders) | 6 (7)
Urinary Frequency (Renal and urinary disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight Decreased (Investigations) | 9 (11)

LIMITATIONS AND CAVEATS:
The primary objective was to determine the number of patients wtih progression-free survival at 6 months. Unfortunately all eligible patients were off therapy before the 6 month time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less